CLINICAL TRIAL: NCT01989260
Title: Effectiveness of Anti-adhesive Gel in Preventing Post Operative Ovarian Adhesions in Women With Pelvic Endometriosis: A Double Blind Randomized Controlled Trial
Brief Title: Post-operative Ovarian Adhesion Study in Women With Endometriosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University College London Hospitals (Other)
Collaborators: Baxter BioScience (Industry)
Responsible Party: Principal Investigator, Katie Pateman, Medical Doctor: Clinical Research Fellow, University College London Hospitals
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Prevention
Other Study IDs: 13/0055; BS12-000796 (Other Grant/Funding Number: Baxter BioScience); 13/LO/0853 (Other: NHS REC)
Record Dates: First submitted 2013-11-14; First posted 2013-11-20 (Estimated); Last update posted 2013-11-20 (Estimated); Status verified 2013-11

CONDITIONS: Endometriosis
Keywords: Endometriosis
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Anti-adhesive gel (Other): An anti-adhesive gel will be administered to one ovary (randomised at the time of laparoscopic surgery to severe endometriosis). The coated ovary will be compared to the non-coated ovary 3 months after surgery to assess for the presence of post-operative ovarian adhesions. Neither the patient nor the person performing the ultrasound scan assessing for the presence of ovarian adhesions will know which was the ovary coated in the anti-adhesive gel.
  Interventions: Device: Anti-adhesive gel

INTERVENTIONS:
Device: Anti-adhesive gel — 4mls of anti-adhesive gel coated to the randomized ovary
  Other Names: Baxter BioScience; CoSeal Surgical Sealant; CE 0123

SUMMARY:
Endometriosis is a common gynaecological condition which typically present with pelvic pain and fertility problems. It is caused by tissues which are similar to the lining of the womb growing inside the women's pelvis. Severe endometriosis is most effectively treated using keyhole surgery. During the operation, endometriosis tissue is removed. However, following successful removal of endometriosis, women may still experience pain because the ovaries sometimes become stuck to the bottom of the pelvis due to post-operative scarring. We want to see if coating one of the ovaries in an anti-scar tissue gel stops the post-operative scarring.

DETAILED DESCRIPTION:
Endometriosis is a common benign condition, affecting women of reproductive age. The disorder is characterized by endometrial surface epithelium, endometrial glands or stroma, found outside the uterus at anatomically ectopic sites.

* Laparoscopic excision of the disease is frequently carried out for the treatment of severe endometriosis. Pelvic adhesions often develop following surgery, restricting the success of treatment. Commercially available anti-adhesive solutions are often used successfully for limiting post-operative adhesions following myomectomy surgery.
* This study aims to assess the effect of resorbable hydrogel anti-adhesive gel following laparoscopic surgery for severe pelvic endometriosis on the prevalence of postoperative ovarian adhesions.
* This is a prospective double blind randomized controlled trial for patients with severe pelvic endometriosis (as defined by the American Society for Reproductive Medicine classification system) requiring extensive laparoscopic dissection (open of one or both para-rectal spaces) with uterine and ovarian preservation.
* Disease severity and eligibility for inclusion into the study will be confirmed at surgery.
* Pre-operatively, all participants will complete a standardized symptom questionnaire detailing the presence and intensity of specific endometriosis symptoms Intra-operatively both ovaries are routinely elevated to the anterior abdominal wall using Prolene suture (ovarian suspension) to facilitate operative access. At the end of the procedure, each participant will be randomized to having only one ovary coated with 4mls of hydrogel anti-adhesive gel, before the ovaries are replaced to their anatomically correct position.
* Three months after surgery, all randomized patients will have a transvaginal ultrasound scan to assess for ovarian mobility and repeat symptom questionnaire.
* Both patients and the person performing the ultrasound scan will be blinded to the randomization process.

ELIGIBILITY:
Inclusion Criteria:

* Women aged between 19-55 years
* diagnosed with severe endometriosis on pre-operative transvaginal ultrasound
* severe endometriosis diagnosed in the surgical context is the opening of one or both para-rectal spaces

Exclusion Criteria:

* inability/unwillingness to provide written consent
* inability to tolerate a transvaginal ultrasound scan
* complications at surgery such as unplanned oophorectomies, bowel injuries or conversion to open surgery

Ages: 19 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2013-12; Primary Completion 2015-04 (Estimated); Study Completion 2015-04 (Estimated)

PRIMARY OUTCOMES:
The prevalence of ovarian adhesions diagnosed by ultrasound after laparoscopic surgery | Ultrasound assessment 3 months post-surgery
  The primary outcome measure is the prevalence of ovarian adhesions diagnosed by ultrasound assessment after surgery. The presence of ovarian adhesions will be assessed by a combination of gentle pressure with the vaginal probe and abdominal pressure with the examiner's free hand as in a bimanual examination. The prevalence of ovarian adhesions will be diagnosed when the ovarian mobility is restricted and the ovary cannot be separated from the peritoneum of the lateral pelvic side wall and/or pouch of Douglas.

SECONDARY OUTCOMES:
The presence, intensity and site of post operative pain | Assessed at 3 months post-operative review

CONTACTS AND LOCATIONS:
Overall Officials: Davor Jurkovic, Study Director — University College London Hospital; Ertan Saridogan, Study Chair — University College London Hospital; Alfred Cutner, Study Chair — University College London Hospital; George Pandis, Study Chair — University College London Hospital
Locations (1):
- University College London Hospital, London, England, United Kingdom